CLINICAL TRIAL: NCT04244812
Title: The Microcirculatory Characteristics of the Heart and Lung Meridians: A Study of CSAP Patients and Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019ZY008-MERIDIAN
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Chronic Stable Angina Pectoris
Keywords: meridians; acupuncture; chronic stable angina pectoris; meridian phenomena
MeSH Terms: interventions — Moxibustion; Laser-Doppler Flowmetry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CSAP group (Other): Participants in the CSAP group will receive examination of laser doppler flowmetry(LDF).
  The LDF probes will be left at 4 measuring acupoints, which include Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan (LU9) and Chize (LU5) of the Lung meridian
  Interventions: Device: Laser doppler flowmetry
- Healthy control group (Other): Participants in the healthy control group will receive examination of laser doppler flowmetry(LDF). The LDF probes will be left at 4 measuring acupoints, which include Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan (LU9) and Chize (LU5) of the Lung meridian.
  Interventions: Device: Laser doppler flowmetry
- Healthy intervention group (Experimental): Participants in the healthy intervention group will receive intervention of moxibustion in the Heart and Lung meridians.
  Interventions: Other: Moxibustion; Device: Laser doppler flowmetry

INTERVENTIONS:
Other: Moxibustion — Two sessions of moxibustion will be performed in the Heart meridian and Lung meridian successively.
  Intervention in the Heart meridian: moxibustion will be performed above Shaohai (HT3) for 15 minutes. During moxibustion, the probes of laser doppler flowmetry will detect the microcirculatory characteristics of three measuring sites, which include the midpoint of the Heart meridian along the left forearm, Chize (LU5) of the Lung meridian, and the midpoint of the Lung meridian along the left forearm.
  Intervention in the Lung meridian: moxibustion will be performed above Chize (LU5) for 15 minutes. During moxibustion, the probes of laser doppler flowmetry will detect the microcirculatory characteristics of three measuring sites, which include the midpoint of the Lung meridian along the left forearm, Shaohai (HT3) of the Heart meridian, and the midpoint of the Heart meridian along the left forearm.
  Arms: Healthy intervention group
Device: Laser doppler flowmetry — Laser doppler flowmetry will be used to detect the microcirculatory characteristics of meridian phenomena

SUMMARY:
This study is designed to detect the microcirculatory characteristics of meridian phenomena by using an objective assessment tool and investigate the site specificity for the meridian-visceral association and surface-surface association between two specific meridians.

DETAILED DESCRIPTION:
The Lung and Heart meridians are chosen as two specific studied meridians. Participants of chronic stable angina pectoris (CSAP) and healthy volunteers will be enrolled.

120 participants will be included and divided into the healthy control group, chronic stable angina pectoris (CSAP) group and healthy intervention group. Laser doppler flowmetry (LDF) will be used to assess the microcirculatory characteristics of meridian phenomena for the Heart and Lung meridians. The site specificity for the meridian-visceral association will be investigated by comparing the microcirculatory difference between the Heart and Lung meridians in the healthy control group and CSAP group. Besides, participants in the healthy intervention group will receive two sessions of moxibustion in the Heart meridian and Lung meridian respectively to explore the site specificity for the surface-surface association.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the CSAP group

* Patients should meet the diagnostic criteria of coronary heart disease, which includes the following items: 1)confirmed old myocardial infarction (MI), or a history of percutaneous coronary intervention(PCI), or coronary artery bypass grafting; 2)50% or more luminal stenosis in at least one coronary artery or major branch segment confirmed by coronary angiogram or CT angiography; 3) myocardial ischemia indicted by exercise stress radionuclide myocardial imaging; 4) treadmill exercise testing is positive (for male patients);
* Patients should meet the diagnostic criteria of CSAP and the Canadian Cardiovascular Society(CCS) classification for CSAP is level II or III;
* The medical history of CSAP is more than 3 months with attacks occurring at least twice weekly in the last month;
* 35 ≤ age ≤75 years, male or female;
* Patients have clear consciousness and could communicate with others normally;
* Patients could understand the full study protocol and written informed consent is signed.

Inclusion criteria for health volunteers

* Healthy volunteers should provide a recent medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
* age≥20 years, male or female;
* Participants have clear consciousness and could communicate with others normally;
* Participants could understand the full study protocol and written informed consent is provided by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for the CSAP group

* Patients with acute coronary syndrome and severe arrhythmias;
* Patients'chest pain is caused by valvular heart disease, hypertrophic cardiomyopathy and dilated cardiomyopathy;
* Patients'chest pain is caused by non-cardiac disease;
* Patients have concomitant conditions of lung diseases, such as obstructive pulmonary disease;
* Patients have serious concomitant conditions and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological and nervous system;
* Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
* Pregnant or lactating patients;
* Patients are participating in other trials.

Exclusion criteria for health volunteers

* Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
* Pregnant or lactating participants ;
* Participants are participating in other trials.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline blood flow curve | 5-minute baseline, 15 minutes during moxibustion and 5 minutes after stopping moxibustion
  Laser doppler flowmetry is used to assess blood flow curve of relevant sites along the Heart and Lung meridians
Change from baseline blood perfusion units | 5-minute baseline, 15 minutes during moxibustion and 5 minutes after stopping moxibustion
  Laser doppler flowmetry is used to assess blood perfusion units of relevant sites along the Heart and Lung meridians

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, M.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

REFERENCES:
- [Background] Hsiu H, Hsu WC, Huang SM, Hsu CL, Lin Wang YY. Spectral analysis of the microcirculatory laser Doppler signal at the Hoku acupuncture point. Lasers Med Sci. 2009 May;24(3):353-8. doi: 10.1007/s10103-008-0569-8. Epub 2008 May 27. PMID 18504639
- [Background] Hsiu H, Hsu WC, Hsu CL, Huang SM, Jan MY, Wang WK, Wang YY. Spectral analysis on the microcirculatory laser Doppler signal at the acupuncture point. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:1084-6. doi: 10.1109/IEMBS.2008.4649348. PMID 19162851
- [Background] Hsiu H, Huang SM, Chao PT, Jan MY, Hsu TL, Wang WK, Wang YY. Microcirculatory characteristics of acupuncture points obtained by laser Doppler flowmetry. Physiol Meas. 2007 Oct;28(10):N77-86. doi: 10.1088/0967-3334/28/10/N01. Epub 2007 Sep 18. PMID 17906382
- [Background] Hsiu H, Hsu WC, Wu YF, Hsu CL, Chen CY. Differences in the skin-surface laser Doppler signals between polycystic ovary syndrome and normal subjects. Microcirculation. 2014 Feb;21(2):124-30. doi: 10.1111/micc.12095. PMID 24118419
- [Derived] Hu H, Jiang Y, Li X, Lou J, Zhang Y, He X, Fang J, Wu Y, Shao X, Fang J. The microcirculatory characteristics of the heart and lung meridians: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Apr;99(14):e19594. doi: 10.1097/MD.0000000000019594. PMID 32243379